CLINICAL TRIAL: NCT05710146
Title: Assessing the Efficacy of Tranexamic Acid (TXA) in Hip Arthroscopy: A Randomized, Controlled Trial
Brief Title: Tranexamic Acid (TXA) in Hip Arthroscopy
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Study was never started. Did not receive funding.
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, Vehniah Tjong, Assistant Professor, Northwestern University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: STU#00215778
Record Dates: First submitted 2022-08-05; First posted 2023-02-02 (Actual); Last update posted 2023-02-02 (Actual); Status verified 2023-01

CONDITIONS: Hip Pain Chronic; Hip Impingement Syndrome; Hip Injuries; Blood Loss; Femoro Acetabular Impingement
Keywords: Hip Arthroscopy; Tranexamic Acid; Intra-operative Blood Loss; Labral Repair of the Hip; Acetabuloplasty
MeSH Terms: conditions — Hip Injuries; Hemorrhage; Femoracetabular Impingement | interventions — Tranexamic Acid; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Tranexamic Acid (Experimental): Patients will be injected with 15 mg/kg of tranexamic acid in 100mL of normal saline via IV access normally established for this procedure.
  Interventions: Drug: Tranexamic acid
- Placebo (Placebo Comparator): Patients will be injected with 100mL of normal saline via IV access normally established for this procedure.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Tranexamic acid — 1 injection of 15mg/kg of TXA in 100mL of normal saline
  Other Names: TXA; Cyklokapron
  Arms: Tranexamic Acid
Drug: Placebo — 1 injection of 100mL of normal saline
  Other Names: normal saline
  Arms: Placebo

SUMMARY:
The primary goal of this study will be to determine if perioperative IV Tranexamic Acid (TXA) administration will reduce intra-operative bleeding and subsequently improve visual clarity during surgery and reduce operative traction time in patients undergoing hip arthroscopy. Additionally, this study aims to determine whether IV TXA injections will reduce post-operative pain and affect hip-specific patient-reported outcomes in patients undergoing hip arthroscopy.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* Scheduled to undergo primary hip arthroscopy for any intra-articular procedure
* Able to complete and understand study materials in English

Exclusion Criteria:

* Age under 18 years
* Cannot complete and understand study materials in English
* Patients undergoing revision surgery
* Patients who have had previous surgery to the study joint
* Patients on drugs that interfere with coagulation or TXA clearance
* Patients with a known allergy to TXA
* Patients with any of the following comorbidities
* Bleeding and/or coagulative disorders
* Renal impairment
* Sickle cell disease
* Thrombotic diseases
* Comorbidities preventing surgery (including pregnancy)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-12 (Estimated); Primary Completion 2024-03 (Estimated); Study Completion 2024-09 (Estimated)

PRIMARY OUTCOMES:
Visual clarity grade | Throughout surgical procedure
  Surgeon-Reported Visual Clarity Grade Grade 1: Active bleeding leading to poor visibility Grade 2: Moderate amount of blood mixed with the irrigation fluid, where the visibility is slightly affected but is acceptable for operating Grade 3: Little or no bleeding; the visibility is excellent to perform the operation

SECONDARY OUTCOMES:
Intra-operative Visibility Score | Throughout surgical procedure
  Number of intra-operative flushes required.
  Scores as follows:
  1. Greater than 13 saline flushes
  2. 8-12 saline flushes
  3. 4-7 saline flushes
  4. 1-3 saline flushes 5 = Zero saline flushes
Operative traction time | Throughout surgical procedure
  Minutes of the procedure in traction
Estimated blood loss | Throughout surgical procedure
  Estimated blood loss during procedure in mL
Post-operative dressing changes | From time of surgery completion through 2 weeks post-op
  Count number of times post-op dressing was changed
Visual Analog Scale (VAS) Pain Score | Pre-operative baseline up through 24 weeks after surgery
  Scored from 0 (no pain) to 10 (worst possible pain)
Complications | From surgery start time through first 6 months post-op
  Number of complications and type of complication will be recorded
Thromboembolic events | From surgery start time through first 6 months post-op
  Number of thromboembolic events
modified Harris Hip Score (mHHS) | Pre-operative baseline up through 24 weeks after surgery
  Subscales regarding pain severity (1 item, 0-44 points), and function (7 items, 0-47 points). Higher overall score corresponds to less disability.
International Hip Outcome Tool 12 (iHOT) | Pre-operative baseline up through 24 weeks after surgery
  12 questions scored from 0 to 100, with 100 being the best function and least amount of symptoms. The final iHOT score equates to the mean of the 12 scores.

CONTACTS AND LOCATIONS:
Overall Officials: Vehniah K Tjong, MD, Principal Investigator — Northwestern Feinberg School of Medicine
Locations (1):
- Northwestern University Feinberg School of Medicine, Chicago, Illinois, United States